CLINICAL TRIAL: NCT00710684
Title: Study AZ3110866, a Fixed Dose Study of SB-742457 Versus Placebo When Added to Existing Donepezil Treatment in Subjects With Mild-to-moderate Alzheimer's Disease
Brief Title: A Study of SB-742457, Added to Donepezil for the Treatment of Mild-to-moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AZ3110866
Record Dates: First submitted 2008-06-30; First posted 2008-07-04 (Estimated); Results first posted 2017-12-07 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-11

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease cognition SB-742457
MeSH Terms: conditions — Alzheimer Disease | interventions — 3-benzenesulfonyl-8-piperazin-1-ylquinoline; Donepezil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- DONEPEZIL + SB-742457 15 MG (Experimental): SB-742457 - 15mg added to existing donepezil treatment
  Interventions: Drug: SB-742457 15mg; Drug: donepezil 5-10mg
- DONEPEZIL + PLACEBO (Placebo Comparator): Placebo added to existing donepezil
  Interventions: Drug: Placebo; Drug: donepezil 5-10mg
- DONEPEZIL + SB-742457 35 MG (Experimental): SB-742457 - 35mg added to existing donepezil
  Interventions: Drug: SB-742457 35mg; Drug: donepezil 5-10mg

INTERVENTIONS:
Drug: SB-742457 15mg — SB-742457 - 15mg added to existing donepezil treatment
  Arms: DONEPEZIL + SB-742457 15 MG
Drug: SB-742457 35mg — SB-742457 - 35mg added to existing donepezil
  Arms: DONEPEZIL + SB-742457 35 MG
Drug: Placebo — Placebo added to existing donepezil
  Arms: DONEPEZIL + PLACEBO
Drug: donepezil 5-10mg — existing donepezil treatment

SUMMARY:
The study is designed to investigate the safety and efficacy of SB-742457 when added to stable donepezil treatment in subjects with mild-to-moderate Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects and their caregivers must provide informed consent prior to study entry.
* Subjects must have a clinical diagnosis of probable mild-to-moderate Alzheimer's disease with no evidence of disorders that are thought to be the cause of, or contributing to the severity of the subject's dementia and a documented history of at least 6 months of ongoing donepezil therapy with stable dosing for at least the last 2 months.
* Subjects must have a regular caregiver who is willing to attend visits, oversee the subject's compliance with the study and report on the subject's status.
* Female subjects of child-bearing potential must agree to abstinence or an approved form of birth control.
* Subjects must have adequate blood pressure and laboratory values.

Exclusion Criteria:

* Subjects with a diagnosis of possible, probable or definite vascular dementia may not participate.
* Subjects with known hypersensitivity to sunlight or a history of seizures, previous exposure to SB-742457, taking agents for which there is a theoretical risk of interaction with SB-742457, or taking medication for Alzheimer's disease or centrally acting agents which might impact study outcomes may not participate.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 682 (Actual)
Dates: Start 2008-07-01 (Actual); Primary Completion 2010-05-21 (Actual); Study Completion 2010-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (88):
- United States (14):
  - GSK Investigational Site, Litchfield Park, Arizona
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Rancho Mirage, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Hallandale, Florida
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Paterson, New Jersey
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Bennington, Vermont
- Argentina (6):
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Ciudad de Buenos Aires, Buenos Aires
  - GSK Investigational Site, La Plata, Buenos Aires
  - GSK Investigational Site, Córdoba, Córdoba Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Santa Fe
- Australia (7):
  - GSK Investigational Site, Kogarah, New South Wales
  - GSK Investigational Site, Herston, Queensland
  - GSK Investigational Site, Woodville, South Australia
  - GSK Investigational Site, Ballarat, Victoria
  - GSK Investigational Site, Heidelberg West, Victoria
  - GSK Investigational Site, Kew, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
- Canada (9):
  - GSK Investigational Site, Saint John, New Brunswick
  - GSK Investigational Site, Kentville, Nova Scotia
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Peterborough, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Greenfield Park, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
  - GSK Investigational Site, Québec
- Chile (3):
  - GSK Investigational Site, Viña del Mar, Región de Valparaíso
  - GSK Investigational Site, Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago
- Czechia (6):
  - GSK Investigational Site, Mělník
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Ostrava
  - GSK Investigational Site, Pardubice
  - GSK Investigational Site, Pilsen
  - GSK Investigational Site, Prague
- Germany (18):
  - GSK Investigational Site, Ellwangen, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Tübingen, Baden-Wurttemberg
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Alzenau in Unterfranken, Bavaria
  - GSK Investigational Site, Günzburg, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Regensburg, Bavaria
  - GSK Investigational Site, Unterhaching, Bavaria
  - GSK Investigational Site, Bad Homburg, Hesse
  - GSK Investigational Site, Achim, Lower Saxony
  - GSK Investigational Site, Schwerin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Aachen, North Rhine-Westphalia
  - GSK Investigational Site, Bad Honnef, North Rhine-Westphalia
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Jena, Thuringia
  - GSK Investigational Site, Berlin
- Italy (15):
  - GSK Investigational Site, Chieti Scalo, Abruzzo
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, San Felice A Cancello - Caserta, Campania
  - GSK Investigational Site, Cassino (FR), Lazio
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Brescia, Lombardy
  - GSK Investigational Site, Castellanza (VA), Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Rho, Lombardy
  - GSK Investigational Site, Turin, Piedmont
  - GSK Investigational Site, Lido Di Camaiore (LU), Tuscany
  - GSK Investigational Site, Pisa, Tuscany
  - GSK Investigational Site, Perugia, Umbria
  - GSK Investigational Site, Valdagno (VI), Veneto
  - GSK Investigational Site, Verona, Veneto
- Spain (10):
  - GSK Investigational Site, Baracaldo/Vizcaya
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Castellon
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, Salamanca
  - GSK Investigational Site, San Sebastián
  - GSK Investigational Site, San Vicente Del Raspeig/Alicante
  - GSK Investigational Site, Valencia

REFERENCES:
- [Derived] Maher-Edwards G, Watson C, Ascher J, Barnett C, Boswell D, Davies J, Fernandez M, Kurz A, Zanetti O, Safirstein B, Schronen JP, Zvartau-Hind M, Gold M. Two randomized controlled trials of SB742457 in mild-to-moderate Alzheimer's disease. Alzheimers Dement (N Y). 2015 May 7;1(1):23-36. doi: 10.1016/j.trci.2015.04.001. eCollection 2015 Jun. PMID 29854923

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 684 participants were randomized from 100 centers i.e. Australia, Argentina, Chile, Canada, United States of America, Czech Republic, Spain, Italy, Germany between 01 July 2008 and 16 November 2010.
Pre-assignment Details: Out of 1132 participants screened, 725 entered into 4-week placebo run-in period out of which 41 participants were placebo run-in failures. Out of 684 participants randomized, 682 were included in safety population (1 participant each from Donepezil+Placebo and Donepezil+SB742457 35 milligram [mg] group failed to take a dose of study medication).
Groups:
- Donepezil + Placebo: Eligible participants who were on donepezil (at least 6 months and a stable regimen for at least 2 months) received placebo tablets matching with SB742457 orally once daily for a treatment period of 48 weeks as an adjunct treatment to stable donepezil therapy. At the end of 24 weeks treatment participants were asked to consent/assent to continue their randomized treatment for a further 24 weeks.
- Donepezil + SB-742457 15 mg: Eligible participants who were on donepezil (at least 6 months and a stable regimen for at least 2 months) received SB742457 15 mg orally once daily for a treatment period of 48 weeks as an adjunct treatment to stable donepezil therapy. At the end of 24 weeks treatment participants were asked to consent/assent to continue their randomized treatment for a further 24 weeks.
- Donepezil + SB-742457 35 mg: Eligible participants who were on donepezil (at least 6 months and a stable regimen for at least 2 months) received SB742457 35 mg orally once daily for a treatment period of 48 weeks as an adjunct treatment to stable donepezil therapy. At the end of 24 weeks treatment participants were asked to consent/assent to continue their randomized treatment for a further 24 weeks.
Period: Overall Study
Arm/Group | Donepezil + Placebo | Donepezil + SB-742457 15 mg | Donepezil + SB-742457 35 mg
Started | 225 | 221 | 236
Completed | 151 | 147 | 172
Not Completed | 74 | 74 | 64
Not completed — Adverse Event | 11 | 19 | 16
Not completed — Lack of Efficacy | 4 | 3 | 5
Not completed — Protocol Violation | 5 | 5 | 5
Not completed — Lost to Follow-up | 4 | 6 | 7
Not completed — Physician Decision | 0 | 2 | 4
Not completed — Withdrawal by Subject | 24 | 18 | 11
Not completed — Missing | 1 | 0 | 0
Not completed — Did not continue after week 24 | 25 | 21 | 16

BASELINE CHARACTERISTICS:
Population: Out of 682 participants, 5 participants did not have at least one post-Baseline or health outcomes assessment. Hence a total of 677 participants were included in intent-to-treat (ITT) population and they were used to assess Baseline characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Donepezil + Placebo | Donepezil + SB-742457 15 mg | Donepezil + SB-742457 35 mg | Total
Number analyzed (Participants) | 223 | 218 | 236 | 677
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.1 (7.49) | 74.2 (6.82) | 73.8 (6.92) | 73.7 (7.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 118 | 148 | 395
  Male | 94 | 100 | 88 | 282
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 2 | 5
  White | 223 | 215 | 233 | 671
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog) Total Score at Week 24
Description: ADAS-cog assessed a range of cognitive abilities including memory, comprehension, orientation in time and place and spontaneous speech. Most items were evaluated by tests, but some were dependent on clinician ratings on a five point scale. There were in all 11 questions. Total scores were calculated as the sum of the individual components. Scores ranged from 0 to 70 with higher scores indicated greater dysfunction. The ADAS-Cog total score was the sum of the calculated scores for questions 1, 2, and 7, and the scores recorded on the case report form (CRF) for questions 3 to 6 and 8 to 11. When a score was missing for one of the questions, the total score was calculated as a weighted average of the scores provided for the remaining ten questions. The change from Baseline was obtained by subtracting the Baseline value from the post-randomization value. Baseline was Week 0 value. Data for adjusted mean is presented.
Time Frame: Baseline(Week 0) and Week 24
Population: ITT population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Donepezil + Placebo | Donepezil + SB-742457 15 mg | Donepezil + SB-742457 35 mg
Number analyzed (Participants) | 193 | 184 | 200
Score on scale | 1.2 (0.45) | 0.5 (0.44) | -0.4 (0.41)
Statistical Analysis 1: Comparison: Donepezil + Placebo vs Donepezil + SB-742457 15 mg; SB-742457 15mg versus placebo at Week 24; Test type: Superiority or Other; p = 0.279, mixed model for repeated measures (MMRM); The MMRM model included fixed categorical terms for treatment, visit, treatment by visit interaction and country; Mean Difference (Net) = -0.7, 95% CI 2-sided [-1.9 to 0.5]
Statistical Analysis 2: Comparison: Donepezil + Placebo vs Donepezil + SB-742457 35 mg; SB-742457 35mg versus placebo at Week 24; Test type: Superiority or Other; p = 0.012, MMRM; The MMRM model included fixed categorical terms for treatment, visit, treatment by visit interaction and country; Mean Difference (Net) = -1.5, 95% CI 2-sided [-2.7 to -0.3]

2. Primary Outcome: Change From Baseline in Clinical Dementia Rating - Sum of Boxes (CDR-SB) Score at Week 24
Description: The CDR-SB is an interviewer administered scale and impairment is scored in each of categories: memory, orientation, judgment and problem solving, community affairs, home and hobbies and personal care. Impairment is scored on a scale in which none = 0, questionable = 0.5, mild = 1, moderate = 2 and severe = 3. The 6 individual category ratings, or "box scores", were added together to give the CDR-Sum of Boxes which ranges from 0-18 (severe impairment). If there were any missing items then CDR-SB was set to missing and was not imputed. The change from Baseline was obtained by subtracting the Baseline value from the post-randomization value. Baseline was Week 0 value. Data for adjusted mean has been presented.
Time Frame: Baseline(Week 0) and Week 24
Population: ITT population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Donepezil + Placebo | Donepezil + SB-742457 15 mg | Donepezil + SB-742457 35 mg
Number analyzed (Participants) | 191 | 184 | 200
Score on scale | 0.9 (0.13) | 0.8 (0.13) | 0.7 (0.11)
Statistical Analysis 1: Comparison: Donepezil + Placebo vs Donepezil + SB-742457 15 mg; SB-742457 15 mg versus placebo at Week 24; Test type: Superiority or Other; p = 0.711, MMRM; The MMRM model included fixed categorical terms for treatment, visit, treatment by visit interaction and country; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.4 to 0.3]
Statistical Analysis 2: Comparison: Donepezil + Placebo vs Donepezil + SB-742457 35 mg; SB-742457 35 mg versus placebo at Week 24; Test type: Superiority or Other; p = 0.462, MMRM; The MMRM model included fixed categorical terms for treatment, visit, treatment by visit interaction and country; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.5 to 0.2]

3. Secondary Outcome: Change From Baseline in Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Total Score at Week 24
Description: RBANS is an individually administered cognitive battery comprising 12 subtests across five domains (Attention, Language, Visuospatial/Constructional Abilities, and Immediate and Delayed memory). Total scores are calculated by adding up the scores for each of the 12 individual subtests and ranges between 0 and 311, where a low score indicates greater impairment. The change from Baseline was obtained by subtracting the Baseline value from the post-randomization value. Baseline was Week 0 value. Data for adjusted mean has been presented.
Time Frame: Baseline (Week 0) and Week 24
Population: ITT population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Donepezil + Placebo | Donepezil + SB-742457 15 mg | Donepezil + SB-742457 35 mg
Number analyzed (Participants) | 190 | 176 | 193
Score on scale | -3.6 (1.18) | -5.9 (1.29) | -4.0 (1.09)
Statistical Analysis 1: Comparison: Donepezil + Placebo vs Donepezil + SB-742457 15 mg; SB-742457 15 mg versus placebo at Week 24; Test type: Superiority or Other; p = 0.174, MMRM; The MMRM model included fixed categorical terms for treatment, visit, treatment by visit interaction and country; Mean Difference (Net) = -2.4, 95% CI 2-sided [-5.8 to 1.1]
Statistical Analysis 2: Comparison: Donepezil + Placebo vs Donepezil + SB-742457 35 mg; SB-742457 35 mg versus placebo at Week 24; Test type: Superiority or Other; p = 0.776, MMRM; The MMRM model included fixed categorical terms for treatment, visit, treatment by visit interaction and country; Mean Difference (Net) = -0.5, 95% CI 2-sided [-3.6 to 2.7]

4. Secondary Outcome: Change From Baseline in ADAS-Cog Total Score at Week 12, 36 and 48
Description: ADAS-cog assessed a range of cognitive abilities including memory, comprehension, orientation in time and place and spontaneous speech. Most items were evaluated by tests, but some were dependent on clinician ratings on a five point scale. There were in all 11 questions. Total scores were calculated as the sum of the individual components. Scores ranged from 0 to 70 with higher scores indicated greater dysfunction. The ADAS-Cog total score was the sum of the calculated scores for questions 1, 2, and 7, and the scores recorded on the CRF for questions 3 to 6 and 8 to 11. In cases where more than one question was missing, a total score was not be imputed. When a score was missing for one of the questions, the total score was calculated as a weighted average of the scores provided for the remaining ten questions. The change from Baseline was obtained by subtracting the Baseline value from the post-randomization value. Baseline was Week 0 value. Data for adjusted mean has been present
Time Frame: Baseline (Week 0) and Week 12, 36 and 48
Population: ITT population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Donepezil + Placebo | Donepezil + SB-742457 15 mg | Donepezil + SB-742457 35 mg
Number analyzed (Participants) | 223 | 218 | 236
Score on scale
  Week 12: number analyzed (Participants) | 206 | 202 | 219
  Week 12 | 0.4 (0.33) | 0.1 (0.37) | -0.9 (0.34)
  Week 36: number analyzed (Participants) | 164 | 156 | 181
  Week 36 | 2.1 (0.45) | 2.1 (0.48) | 0.9 (0.45)
  Week 48: number analyzed (Participants) | 145 | 142 | 170
  Week 48 | 3.4 (0.52) | 3.4 (0.60) | 1.8 (0.50)
Statistical Analysis 1: Comparison: Donepezil + Placebo vs Donepezil + SB-742457 15 mg; SB-742457 15 mg versus placebo at Week 12; Test type: Superiority or Other; p = 0.631, MMRM; The MMRM model included fixed categorical terms for treatment, visit, treatment by visit interaction and country; Mean Difference (Net) = -0.2, 95% CI 2-sided [-1.2 to 0.7]
Statistical Analysis 2: Comparison: Donepezil + Placebo vs Donepezil + SB-742457 35 mg; SB-742457 35 mg versus placebo at Week 12; Test type: Superiority or Other; p = 0.006, MMRM; The MMRM model included fixed categorical terms for treatment, visit, treatment by visit interaction and country; Mean Difference (Net) = -1.3, 95% CI 2-sided [-2.2 to -0.4]
Statistical Analysis 3: Comparison: Donepezil + Placebo vs Donepezil + SB-742457 15 mg; SB-742457 15 mg versus placebo at Week 36; Test type: Superiority or Other; p = 0.947, MMRM; The MMRM model included fixed categorical terms for treatment, visit, treatment by visit interaction and country; Mean Difference (Net) = 0.0, 95% CI 2-sided [-1.3 to 1.2]
Statistical Analysis 4: Comparison: Donepezil + Placebo vs Donepezil + SB-742457 35 mg; SB-742457 35 mg versus placebo at Week 36; Test type: Superiority or Other; p = 0.057, MMRM; The MMRM model included fixed categorical terms for treatment, visit, treatment by visit interaction and country; Mean Difference (Net) = -1.2, 95% CI 2-sided [-2.5 to 0.0]
Statistical Analysis 5: Comparison: Donepezil + Placebo vs Donepezil + SB-742457 15 mg; SB-742457 15 mg versus placebo at Week 48; Test type: Superiority or Other; p = 0.925, MMRM; The MMRM model included fixed categorical terms for treatment, visit, treatment by visit interaction and country; Mean Difference (Net) = -0.1, 95% CI 2-sided [-1.6 to 1.5]
Statistical Analysis 6: Comparison: Donepezil + Placebo vs Donepezil + SB-742457 35 mg; SB-742457 35 mg versus placebo at Week 48; Test type: Superiority or Other; p = 0.024, MMRM; The MMRM model included fixed categorical terms for treatment, visit, treatment by visit interaction and country; Mean Difference (Net) = -1.6, 95% CI 2-sided [-3.1 to -0.2]

5. Secondary Outcome: Change From Baseline in CDR-SB Score at Week 12, 36 and 48
Description: as for outcome 2
Time Frame: Baseline (Week 0) and Week 12, 36, 48
Population: ITT population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Donepezil + Placebo | Donepezil + SB-742457 15 mg | Donepezil + SB-742457 35 mg
Number analyzed (Participants) | 223 | 218 | 236
Score on scale
  Week 12: number analyzed (Participants) | 203 | 199 | 221
  Week 12 | 0.5 (0.10) | 0.4 (0.09) | 0.2 (0.08)
  Week 36: number analyzed (Participants) | 163 | 154 | 179
  Week 36 | 1.2 (0.15) | 1.4 (0.18) | 1.0 (0.13)
  Week 48: number analyzed (Participants) | 146 | 142 | 170
  Week 48 | 1.6 (0.16) | 1.9 (0.20) | 1.5 (0.16)
Statistical Analysis 1: Comparison: Donepezil + Placebo vs Donepezil + SB-742457 15 mg; SB-742457 15 mg versus placebo at Week 12; Test type: Superiority or Other; p = 0.387, MMRM; The MMRM model included fixed categorical terms for treatment, visit, treatment by visit interaction and country; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.4 to 0.1]
Statistical Analysis 2: Comparison: Donepezil + Placebo vs Donepezil + SB-742457 35 mg; SB-742457 35 mg versus placebo at Week 12; Test type: Superiority or Other; p = 0.018, MMRM; Mean Difference (Net) = -0.3, 95% CI 2-sided [-0.5 to -0.1]
Statistical Analysis 3: Comparison: Donepezil + Placebo vs Donepezil + SB-742457 15 mg; SB-742457 15 mg versus placebo at Week 36; Test type: Superiority or Other; p = 0.439, MMRM; The MMRM model included fixed categorical terms for treatment, visit, treatment by visit interaction and country; Mean Difference (Net) = 0.2, 95% CI 2-sided [-0.3 to 0.6]
Statistical Analysis 4: Comparison: Donepezil + Placebo vs Donepezil + SB-742457 35 mg; SB-742457 35 mg versus placebo at Week 36; Test type: Superiority or Other; p = 0.336, MMRM; The MMRM model included fixed categorical terms for treatment, visit, treatment by visit interaction and country; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.6 to 0.2]
Statistical Analysis 5: Comparison: Donepezil + Placebo vs Donepezil + SB-742457 15 mg; SB-742457 15 mg versus placebo at Week 48; Test type: Superiority or Other; p = 0.190, MMRM; The MMRM model included fixed categorical terms for treatment, visit, treatment by visit interaction and country; Mean Difference (Net) = 0.3, 95% CI 2-sided [-0.2 to 0.8]
Statistical Analysis 6: Comparison: Donepezil + Placebo vs Donepezil + SB-742457 35 mg; SB-742457 35 mg versus placebo at Week 48; Test type: Superiority or Other; p = 0.787, MMRM; The MMRM model included fixed categorical terms for treatment, visit, treatment by visit interaction and country; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.5 to 0.4]

6. Secondary Outcome: Change From Baseline in RBANS Score at Week 12, 36 and 48
Description: as for outcome 3
Time Frame: Baseline (Week 0) and Week 12, 36 and 48
Population: ITT population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Donepezil + Placebo | Donepezil + SB-742457 15 mg | Donepezil + SB-742457 35 mg
Number analyzed (Participants) | 223 | 218 | 236
Score on scale
  Week 12: number analyzed (Participants) | 200 | 194 | 214
  Week 12 | -7.2 (0.94) | -8.5 (1.02) | -6.5 (0.79)
  Week 36: number analyzed (Participants) | 161 | 153 | 174
  Week 36 | -3.9 (1.32) | -4.8 (1.21) | -1.8 (1.19)
  Week 48: number analyzed (Participants) | 143 | 136 | 164
  Week 48 | -7.3 (1.36) | -9.4 (1.45) | -4.7 (1.25)
Statistical Analysis 1: Comparison: Donepezil + Placebo vs Donepezil + SB-742457 15 mg; SB-742457 15 mg versus placebo at Week 12; Test type: Superiority or Other; p = 0.337, MMRM; The MMRM model included fixed categorical terms for treatment, visit, treatment by visit interaction and country; Mean Difference (Net) = -1.3, 95% CI 2-sided [-4.0 to 1.4]
Statistical Analysis 2: Comparison: Donepezil + Placebo vs Donepezil + SB-742457 35 mg; SB-742457 35 mg versus placebo at Week 12; Test type: Superiority or Other; p = 0.596, MMRM; The MMRM model included fixed categorical terms for treatment, visit, treatment by visit interaction and country; Mean Difference (Net) = 0.6, 95% CI 2-sided [-1.7 to 3.0]
Statistical Analysis 3: Comparison: Donepezil + Placebo vs Donepezil + SB-742457 15 mg; SB-742457 15 mg versus placebo at Week 36; Test type: Superiority or Other; p = 0.634, MMRM; The MMRM model included fixed categorical terms for treatment, visit, treatment by visit interaction and country; Mean Difference (Net) = -0.9, 95% CI 2-sided [-4.4 to 2.7]
Statistical Analysis 4: Comparison: Donepezil + Placebo vs Donepezil + SB-742457 35 mg; SB-742457 35 mg versus placebo at Week 36; Test type: Superiority or Other; p = 0.238, MMRM; The MMRM model included fixed categorical terms for treatment, visit, treatment by visit interaction and country; Mean Difference (Net) = 2.1, 95% CI 2-sided [-1.4 to 5.6]
Statistical Analysis 5: Comparison: Donepezil + Placebo vs Donepezil + SB-742457 15 mg vs Donepezil + SB-742457 35 mg; SB-742457 15 mg versus placebo at Week 48; Test type: Superiority or Other; p = 0.292, MMRM; The MMRM model included fixed categorical terms for treatment, visit, treatment by visit interaction and country; Mean Difference (Net) = -2.1, 95% CI 2-sided [-6.0 to 1.8]
Statistical Analysis 6: Comparison: Donepezil + Placebo vs Donepezil + SB-742457 35 mg; SB-742457 35 mg versus placebo at Week 48; Test type: Superiority or Other; p = 0.161, MMRM; The MMRM model included fixed categorical terms for treatment, visit, treatment by visit interaction and country; Mean Difference (Net) = 2.6, 95% CI 2-sided [-1.0 to 6.2]

7. Secondary Outcome: Change From Baseline in Alzheimer's Disease Co-operative Study Group - Activities of Daily Living Inventory (ADCS- ADL) Total Score at Weeks 12, 24, 36 and 48
Description: The ADCS-ADL is an interviewer-administered informant-based scale where the informant (caregiver) responds to 23 activities of daily living questions about the participant. The questions ranged from basic to instrumental activities of daily living and take approximately 20 minutes to complete. The Total score ranges from 0-78 and a higher score signified greater functional ability. The questionnaire was split into two types of questions, an initial question relating to whether a participant had completed a particular activity and then a follow on question which scored how much assistance the participant had required if they had performed that particular activity. The total score was calculated by adding up the responses for each of the individual activities. The change from Baseline was obtained by subtracting the Baseline value from the post-randomization value. Baseline was Week 0 value. Data for adjusted mean has been presented.
Time Frame: Baseline (Week 0) and Week 12, 24, 36 and 48
Population: ITT population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Donepezil + Placebo | Donepezil + SB-742457 15 mg | Donepezil + SB-742457 35 mg
Number analyzed (Participants) | 223 | 218 | 236
Score on scale
  Week 12: number analyzed (Participants) | 202 | 200 | 222
  Week 12 | -1.4 (0.57) | -0.8 (0.49) | 0.3 (0.47)
  Week 24: number analyzed (Participants) | 192 | 185 | 209
  Week 24 | -3.4 (0.66) | -1.9 (0.61) | -1.4 (0.60)
  Week 36: number analyzed (Participants) | 164 | 159 | 183
  Week 36 | -3.7 (0.67) | -3.8 (0.80) | -1.8 (0.65)
  Week 48: number analyzed (Participants) | 147 | 144 | 171
  Week 48 | -5.5 (0.85) | -5.0 (0.87) | -3.5 (0.76)
Statistical Analysis 1: Comparison: Donepezil + Placebo vs Donepezil + SB-742457 15 mg; SB-742457 15 mg versus placebo at Week 12; Test type: Superiority or Other; p = 0.396, MMRM; The MMRM model included fixed categorical terms for treatment, visit, treatment by visit interaction and country; Mean Difference (Net) = 0.6, 95% CI 2-sided [-0.8 to 2.1]
Statistical Analysis 2: Comparison: Donepezil + Placebo vs Donepezil + SB-742457 35 mg; SB-742457 35 mg versus placebo at Week 12; Test type: Superiority or Other; p = 0.019, MMRM; The MMRM model included fixed categorical terms for treatment, visit, treatment by visit interaction and country; Mean Difference (Net) = 1.7, 95% CI 2-sided [0.3 to 3.2]
Statistical Analysis 3: Comparison: Donepezil + Placebo vs Donepezil + SB-742457 15 mg; SB-742457 15 mg versus placebo at Week 24; Test type: Superiority or Other; p = 0.110, MMRM; The MMRM model included fixed categorical terms for treatment, visit, treatment by visit interaction and country; Mean Difference (Net) = 1.4, 95% CI 2-sided [-0.3 to 3.2]
Statistical Analysis 4: Comparison: Donepezil + Placebo vs Donepezil + SB-742457 35 mg; SB-742457 35 mg versus placebo at Week 24; Test type: Superiority or Other; p = 0.024, MMRM; The MMRM model included fixed categorical terms for treatment, visit, treatment by visit interaction and country; Mean Difference (Net) = 2.0, 95% CI 2-sided [0.3 to 3.7]
Statistical Analysis 5: Comparison: Donepezil + Placebo vs Donepezil + SB-742457 15 mg; SB-742457 15 mg versus placebo ate Week 36; Test type: Superiority or Other; p = 0.944, MMRM; The MMRM model included fixed categorical terms for treatment, visit, treatment by visit interaction and country; Mean Difference (Net) = -0.1, 95% CI 2-sided [-2.1 to 2.0]
Statistical Analysis 6: Comparison: Donepezil + Placebo vs Donepezil + SB-742457 35 mg; SB-742457 35 mg versus placebo at Week 36; Test type: Superiority or Other; p = 0.037, MMRM; The MMRM model included fixed categorical terms for treatment, visit, treatment by visit interaction and country; Mean Difference (Net) = 1.9, 95% CI 2-sided [0.1 to 3.8]
Statistical Analysis 7: Comparison: Donepezil + Placebo vs Donepezil + SB-742457 15 mg; SB-742457 15 mg versus placebo at Week 48; Test type: Superiority or Other; p = 0.705, MMRM; The MMRM model included fixed categorical terms for treatment, visit, treatment by visit interaction and country; Mean Difference (Net) = 0.5, 95% CI 2-sided [-1.9 to 2.9]
Statistical Analysis 8: Comparison: Donepezil + Placebo vs Donepezil + SB-742457 35 mg; SB-742457 35 mg versus placebo at Week 48; Test type: Superiority or Other; p = 0.088, MMRM; The MMRM model included fixed categorical terms for treatment, visit, treatment by visit interaction and country; Mean Difference (Net) = 1.9, 95% CI 2-sided [-0.3 to 4.2]

8. Secondary Outcome: Change From Baseline in Mini Mental State Examination (MMSE) Total Score at Week 24 and 48
Description: The MMSE consisted of 11 items covering orientation, memory (recent and immediate), concentration, language and praxis. Scores ranged from 0 to 30, with lower scores indicating greater cognitive impairment. Scores for each of the 11 individual tests were not recorded on the CRF, therefore if any item was missing then the total score was be set to missing. The change from Baseline was obtained by subtracting the Baseline value from the post-randomization value. Baseline was Week 0 value. Data for adjusted mean has been presented.
Time Frame: Baseline (Week 0) and Week 24 and 48
Population: ITT population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Donepezil + Placebo | Donepezil + SB-742457 15 mg | Donepezil + SB-742457 35 mg
Number analyzed (Participants) | 223 | 218 | 236
Score on scale
  Week 24: number analyzed (Participants) | 196 | 188 | 209
  Week 24 | -0.4 (0.21) | -0.3 (0.23) | 0.1 (0.21)
  Week 48: number analyzed (Participants) | 149 | 145 | 172
  Week 48 | -1.1 (0.28) | -1.3 (0.33) | -0.7 (0.27)
Statistical Analysis 1: Comparison: Donepezil + Placebo vs Donepezil + SB-742457 15 mg; SB-742457 15 mg versus placebo at Week 24; Test type: Superiority or Other; p = 0.962, MMRM; The MMRM model included fixed categorical terms for treatment, visit, treatment by visit interaction and country; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.6 to 0.6]
Statistical Analysis 2: Comparison: Donepezil + Placebo vs Donepezil + SB-742457 35 mg; SB-742457 35 mg versus placebo at Week 24; Test type: Superiority or Other; p = 0.134, MMRM; The MMRM model included fixed categorical terms for treatment, visit, treatment by visit interaction and country; Mean Difference (Net) = 0.4, 95% CI 2-sided [-0.1 to 1.0]
Statistical Analysis 3: Comparison: Donepezil + Placebo vs Donepezil + SB-742457 15 mg; SB-742457 15 mg versus placebo at Week 48; Test type: Superiority or Other; p = 0.782, MMRM; The MMRM model included fixed categorical terms for treatment, visit, treatment by visit interaction and country; Mean Difference (Net) = -0.1, 95% CI 2-sided [-1.0 to 0.7]
Statistical Analysis 4: Comparison: Donepezil + Placebo vs Donepezil + SB-742457 35 mg; SB-742457 35 mg versus placebo at Week 48; Test type: Superiority or Other; p = 0.268, MMRM; The MMRM model included fixed categorical terms for treatment, visit, treatment by visit interaction and country; Mean Difference (Net) = 0.4, 95% CI 2-sided [-0.3 to 1.2]

9. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) During Treatment Phase
Description: An AE was defined as any untoward medical occurrence that occurred during the course of the trial after study treatment had started. An adverse event was therefore any unfavorable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. An SAE was any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity, and congenital anomaly/birth defect.
Time Frame: Up to follow-up i.e. 2 weeks post end of treatment (Week 24, Week 48 or Early Withdrawal)
Population: Safety population consisted of all participants randomized to treatment who had received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Donepezil + Placebo | Donepezil + SB-742457 15 mg | Donepezil + SB-742457 35 mg
Number analyzed (Participants) | 225 | 221 | 236
Participants
  Any AE | 125 | 137 | 146
  Any SAE | 17 | 26 | 27

10. Secondary Outcome: Number of Participants With Parameters of Clinical Concern - Hematology
Description: Only parameters with values have been presented. Data has been reported for number of participants with high and/ or low values for Eosinophils (high-2), Hematocrit (low- 0.8, high-1.2), Lymphocytes (low-0.75, high-1.5), Mean Corpuscle Hemoglobin (MCH) (low-0.8, high-1.2), Monocytes(low-0.75, high-2), Neutrophil bands (high-10), Platelet count (low-100, high-500), Segmented Neutrophils (low-0.75, high-1.3), Total Neutrophils (low-0.75, high-1.5), and white blood cells (WBC) (low-3, high-15).
Time Frame: Up to Week 48
Population: Safety population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Donepezil + Placebo | Donepezil + SB-742457 15 mg | Donepezil + SB-742457 35 mg
Number analyzed (Participants) | 225 | 221 | 236
Participants
  Eosinophils, high: number analyzed (Participants) | 222 | 217 | 235
  Eosinophils, high | 1 | 0 | 4
  Hematocrit, low: number analyzed (Participants) | 222 | 217 | 235
  Hematocrit, low | 2 | 2 | 1
  Hematocrit, high: number analyzed (Participants) | 222 | 217 | 235
  Hematocrit, high | 0 | 1 | 0
  Hemoglobin, low: number analyzed (Participants) | 222 | 217 | 235
  Hemoglobin, low | 5 | 3 | 8
  Hemoglobin, high: number analyzed (Participants) | 222 | 217 | 235
  Hemoglobin, high | 3 | 1 | 0
  Lymphocytes, low: number analyzed (Participants) | 222 | 217 | 235
  Lymphocytes, low | 6 | 5 | 7
  Lymphocytes, high: number analyzed (Participants) | 222 | 217 | 235
  Lymphocytes, high | 0 | 2 | 1
  MCH, low: number analyzed (Participants) | 204 | 198 | 216
  MCH, low | 0 | 1 | 0
  MCV, low: number analyzed (Participants) | 222 | 217 | 235
  MCV, low | 0 | 1 | 0
  Monocytes, low: number analyzed (Participants) | 222 | 217 | 235
  Monocytes, low | 35 | 32 | 32
  Monocytes, high: number analyzed (Participants) | 222 | 217 | 235
  Monocytes, high | 0 | 1 | 0
  Neutrophil bands, high: number analyzed (Participants) | 1 | 3 | 3
  Neutrophil bands, high | 0 | 1 | 1
  Platelet count, low: number analyzed (Participants) | 222 | 216 | 235
  Platelet count, low | 1 | 4 | 3
  Platelet count, high: number analyzed (Participants) | 222 | 216 | 235
  Platelet count, high | 2 | 3 | 5
  Segmented Neutrophils, low: number analyzed (Participants) | 222 | 217 | 235
  Segmented Neutrophils, low | 7 | 3 | 7
  Segmented Neutrophils, high: number analyzed (Participants) | 222 | 217 | 235
  Segmented Neutrophils, high | 3 | 4 | 5
  Total Neutrophils, low: number analyzed (Participants) | 222 | 217 | 235
  Total Neutrophils, low | 7 | 3 | 7
  Total Neutrophils, high: number analyzed (Participants) | 222 | 217 | 235
  Total Neutrophils, high | 0 | 3 | 2
  WBC, low: number analyzed (Participants) | 222 | 217 | 235
  WBC, low | 4 | 1 | 5
  WBC, high: number analyzed (Participants) | 222 | 217 | 235
  WBC, high | 0 | 3 | 2

11. Secondary Outcome: Number of Participants With Parameters of Clinical Concern - Clinical Chemistry
Description: Only parameters with values have been presented. Data has been reported for number of participants with high and/ or low values for Alanine Amino Transferase (ALT) (high-1.5), Alkaline Phosphatase (high-1.5), Aspartate Amino Transferase (ASAT) (high-1.5), BUN/Creatinine ratio (high-1.5), Calcium (low- 0.75, high-1.25), Carbon dioxide content/Bicarbonate (low-15, high- 40), Cholesterol (high-1.25), Creatine Kinase ((low- 0.5, high-1.25), Creatinine (low- 0.5, high-1.25), Direct Bilirubin (high-1.5), Gamma Glutamyl Transferase (GGT) (high-2), Glucose (low- 3.6, high-7.8), HDL Cholesterol (low-0.65), LDL Cholesterol (hig-1.25), Magnesium (low-0.5, high-2), Phosphorus inorganic (low- 0.5, high-1.5), Potassium (low- 3, high-5.5), Sodium (low- 130, high-150), Total Bilirubin (high-1.5), Triglycerides (high -4) and Urea/BUN (high-11).
Time Frame: Up to Week 48
Population: Safety population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Donepezil + Placebo | Donepezil + SB-742457 15 mg | Donepezil + SB-742457 35 mg
Number analyzed (Participants) | 225 | 221 | 236
Participants
  ALT, high: number analyzed (Participants) | 222 | 217 | 235
  ALT, high | 2 | 4 | 4
  Alkaline Phosphatase, high: number analyzed (Participants) | 222 | 217 | 235
  Alkaline Phosphatase, high | 5 | 6 | 4
  ASAT, high: number analyzed (Participants) | 222 | 217 | 235
  ASAT, high | 2 | 7 | 4
  BUN/Creatinine ratio, high: number analyzed (Participants) | 222 | 217 | 235
  BUN/Creatinine ratio, high | 11 | 7 | 5
  Calcium, low: number analyzed (Participants) | 222 | 217 | 235
  Calcium, low | 0 | 0 | 1
  Carbon dioxide content/Bicarbonate, low: number analyzed (Participants) | 222 | 217 | 235
  Carbon dioxide content/Bicarbonate, low | 3 | 2 | 2
  Cholesterol, high: number analyzed (Participants) | 204 | 196 | 215
  Cholesterol, high | 11 | 4 | 7
  Creatine Kinase, high: number analyzed (Participants) | 204 | 196 | 215
  Creatine Kinase, high | 5 | 2 | 6
  Creatinine, high: number analyzed (Participants) | 222 | 217 | 235
  Creatinine, high | 3 | 3 | 5
  Direct Bilirubin, high: number analyzed (Participants) | 222 | 217 | 235
  Direct Bilirubin, high | 2 | 1 | 1
  GGT, high: number analyzed (Participants) | 222 | 217 | 235
  GGT, high | 5 | 7 | 7
  Glucose, low: number analyzed (Participants) | 222 | 217 | 235
  Glucose, low | 17 | 24 | 13
  Glucose, high: number analyzed (Participants) | 222 | 217 | 235
  Glucose, high | 54 | 42 | 54
  HDL Cholesterol, direct, low: number analyzed (Participants) | 204 | 195 | 215
  HDL Cholesterol, direct, low | 3 | 0 | 2
  LDL Cholesterol, high: number analyzed (Participants) | 201 | 195 | 214
  LDL Cholesterol, high | 35 | 29 | 40
  Magnesium, low: number analyzed (Participants) | 204 | 195 | 215
  Magnesium, low | 0 | 1 | 0
  Phosphorus, inorganic, high: number analyzed (Participants) | 204 | 196 | 215
  Phosphorus, inorganic, high | 0 | 0 | 1
  Potassium, high: number analyzed (Participants) | 222 | 217 | 235
  Potassium, high | 2 | 10 | 9
  Sodium, high: number analyzed (Participants) | 222 | 217 | 235
  Sodium, high | 0 | 1 | 1
  Total Bilirubin, high: number analyzed (Participants) | 222 | 217 | 235
  Total Bilirubin, high | 2 | 1 | 1
  Triglycerides, high: number analyzed (Participants) | 204 | 196 | 215
  Triglycerides, high | 1 | 0 | 0
  Urea/BUN, high: number analyzed (Participants) | 222 | 217 | 235
  Urea/BUN, high | 17 | 12 | 25

12. Secondary Outcome: Exposure Estimates for SB-742457 : Area Under the Concentration Time Curve Over the Dosing Interval at Steady State (AUCτss)
Description: AUCτss of SB-742457 was estimated via nonlinear mixed effect analysis. This pharmacokinetic(PK) model was a steady state one compartment model with first-order absorption, with between participant variability on clearance and volume of distribution.
Time Frame: Post-dose at 3, 8 and 24 hours on Week 0, 1, 3, 6, 12, 18, 24, 30, 36, 42 and 48
Population: PK population included all participants for whom a pharmacokinetic sample was obtained and analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram hour per milliliter (ng*h/mL)
Arm/Group | Donepezil + SB-742457 15 mg | Donepezil + SB-742457 35 mg
Number analyzed (Participants) | 215 | 233
Nanogram hour per milliliter (ng*h/mL) | 1640.76 (35.96) | 4160.29 (31.67)

13. Secondary Outcome: Exposure Estimates for SB-742457 : Minimum Concentrations at Steady State (Cmin-ss)
Description: Cmin-ss was estimated via nonlinear mixed effect analysis. This PK model was a steady state one compartment model with first-order absorption, with between participant variability on clearance and volume of distribution.
Time Frame: Post-dose at 3, 8 and 24 hours on Week 0, 1, 3, 6, 12, 18, 24, 30, 36, 42 and 48
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Donepezil + SB-742457 15 mg | Donepezil + SB-742457 35 mg
Number analyzed (Participants) | 215 | 233
ng/mL | 53.42 (38.58) | 135.05 (33.08)

14. Secondary Outcome: Exposure Estimates for Donepezil (Cavgss)
Description: Participants who were on donepezil (at least 6 months and a stable regimen for at least 2 months) were allowed to participate in this study. Cavgss for donepezil approximately 12 to 20 hours after dosing were summarized by donepezil dose level 5 mg/7.5 mg/10 mg/15 mg.
Time Frame: Post-dose at 12 to 20 hours on Week 0, 1, 3, 6, 12, 18, 24, 30, 36, 42 and 48
Population: Donepezil PK population comprised of participants who received a stable dose of donepezil 5 mg/7.5 mg/10 mg/15 mg. Analysis is exclusively for Cavgss of donepezil therefore the two arms SB-742457 15 mg and SB-742457 35 mg have not been presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Donepezil 5 mg: Participants received a stable dose of donepezil 5 mg at least for 6 months and a stable regimen for at least 2 months. The participants received SB742457 15 mg or 35 mg or placebo matching with SB742457 orally once daily for a treatment period of 48 weeks as an adjunct treatment to stable donepezil therapy.
- Donepezil 7.5 mg: Participants received a stable dose of donepezil 7.5 mg at least for 6 months and a stable regimen for at least 2 months. The participants received SB742457 15 mg or 35 mg or placebo matching with SB742457 orally once daily for a treatment period of 48 weeks as an adjunct treatment to stable donepezil therapy.
- Donepezil 10 mg: Participants received a stable dose of donepezil 10 mg at least for 6 months and a stable regimen for at least 2 months. The participants received SB742457 15 mg or 35 mg or placebo matching with SB742457 orally once daily for a treatment period of 48 weeks as an adjunct treatment to stable donepezil therapy.
- Donepezil 15 mg: Participants received a stable dose of donepezil 15 mg at least for 6 months and a stable regimen for at least 2 months. The participants received SB742457 15 mg or 35 mg or placebo matching with SB742457 orally once daily for a treatment period of 48 weeks as an adjunct treatment to stable donepezil therapy.
Arm/Group | Donepezil 5 mg | Donepezil 7.5 mg | Donepezil 10 mg | Donepezil 15 mg
Number analyzed (Participants) | 179 | 1 | 484 | 1
ng/mL | 20.72 (45.07) | 17.68 (NA) — Only one participant was analyzed, hence, dispersion value could not be generated. | 39.79 (46.62) | 36.60 (NA) — Only one participant was analyzed.

15. Secondary Outcome: Change From Baseline in ADAS-Cog Scale in Participants With APOE4 Gene
Description: Genetic analyses was conducted to assess the effect of APOE4 carriage. ADAS-cog assessed a range of cognitive abilities including memory, comprehension, orientation in time and place and spontaneous speech. Most items were evaluated by tests, but some were dependent on clinician ratings on a five-point scale. There were in all 11 questions. Total scores were calculated as the sum of the individual components. Scores ranged from 0 to 70 with higher scores indicating greater dysfunction. The ADAS-Cog total score was the sum of the calculated scores for questions 1, 2, and 7, and the scores were recorded on the CRF for questions 3 to 6 and 8 to 11. When a score was missing for one of the questions, the total score was calculated as a weighted average of the scores provided for the remaining ten questions. Baseline was Week 0 value. The change from Baseline was obtained by subtracting the Baseline value from the post-randomization value.
Time Frame: Baseline (Week 0) to Week 24 and Week 48
Population: PGx ITT Population consisted of all participants in the ITT population who had evaluable PGx data. Only those participants with APOE gene and available at the specified time point were analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Donepezil + Placebo | Donepezil + SB-742457 15 mg | Donepezil + SB-742457 35 mg
Number analyzed (Participants) | 206 | 202 | 219
Score on scale
  Week 24: number analyzed (Participants) | 98 | 94 | 114
  Week 24 | 1.9 (5.58) | 1.0 (6.63) | -0.1 (5.40)
  Week 48: number analyzed (Participants) | 74 | 72 | 90
  Week 48 | 4.7 (6.52) | 4.2 (7.46) | 1.8 (5.72)

16. Secondary Outcome: Change From Baseline in CDR-SB Scale in Participants With APOE4 Gene
Description: Genetic analyses was conducted to assess the effect of APOE4 carriage. The CDR-SB is an interviewer administered scale and impairment is scored in following categories: memory, orientation, judgment and problem solving, community affairs, home and hobbies and personal care. Impairment was scored on a scale in which none =0, questionable =0.5, mild =1, moderate =2 and severe =3. The 6 individual category ratings, or "box scores", were added together to give the CDR-Sum of Boxes which ranges from 0-18, with higher score indicating severe impairment. If there were any missing items then CDR-SB was set to missing and was not imputed. Baseline was Week 0 value. The change from Baseline was obtained by subtracting the Baseline value from the post-randomization value.
Time Frame: Baseline (Week 0) to Week 24 and Week 48
Population: PGx ITT Population. Only those participants with APOE gene and available at the specified time point were analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Donepezil + Placebo | Donepezil + SB-742457 15 mg | Donepezil + SB-742457 35 mg
Number analyzed (Participants) | 206 | 202 | 219
Score on scale
  Week 24: number analyzed (Participants) | 95 | 94 | 113
  Week 24 | 1.1 (2.02) | 0.6 (1.59) | 0.8 (1.47)
  Week 48: number analyzed (Participants) | 75 | 71 | 91
  Week 48 | 1.8 (1.98) | 1.5 (2.11) | 1.4 (1.92)

17. Secondary Outcome: Change From Baseline in RBANS Scale in Participants With APOE4 Gene
Description: Genetic analyses was conducted to assess the effect of APOE4 carriage. RBANS is an individually administered cognitive battery comprising 12 subtests across five domains (Attention, Language, Visuospatial/Constructional Abilities, and Immediate and Delayed memory). Total scores are calculated by adding up the scores for each of the 12 individual subtests and ranges between 0 and 311, where a low score indicates greater impairment. Baseline was Week 0 value. The change from Baseline was obtained by subtracting the Baseline value from the post-randomization value.
Time Frame: Baseline (Week 0) to Week 24 and Week 48
Population: PGx ITT Population. Only those participants with APOE gene and available at the specified time point were analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Donepezil + Placebo | Donepezil + SB-742457 15 mg | Donepezil + SB-742457 35 mg
Number analyzed (Participants) | 206 | 202 | 219
Score on scale
  Week 24: number analyzed (Participants) | 96 | 94 | 110
  Week 24 | -5.2 (14.30) | -6.0 (20.07) | -6.0 (14.84)
  Week 48: number analyzed (Participants) | 74 | 72 | 87
  Week 48 | -7.7 (16.46) | -11.3 (16.13) | -5.9 (14.04)

ADVERSE EVENTS:
Time Frame: AE data was collected up to follow-up i.e. 2 weeks post end of treatment Up to follow-up i.e. 2 weeks post end of treatment (Week 24, Week 48 or Early Withdrawal).
Description: Safety population consisted of all participants randomized to treatment who had received at least one dose of study medication. Safety population was used for the analysis of SAE and nSAE.
Arm/Group | Donepezil + Placebo | Donepezil + SB-742457 15 mg | Donepezil + SB-742457 35 mg
All-Cause Mortality (participants affected / at risk) | 1/225 | 5/221 | 4/236
Serious Adverse Events (participants affected / at risk) | 17/225 | 26/221 | 27/236
Other Adverse Events (participants affected / at risk) | 41/225 | 32/221 | 33/236
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Donepezil + Placebo (N=225) | Donepezil + SB-742457 15 mg (N=221) | Donepezil + SB-742457 35 mg (N=236)
Cerebrovascular accident (Nervous system disorders) | 1 | 3 | 1
Syncope (Nervous system disorders) | 1 | 1 | 2
Cerebral haemorrhage (Nervous system disorders) | 0 | 2 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0
Dementia Alzheimer's type (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Psychomotor hyperactivity (Nervous system disorders) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 3 | 1 | 3
Urinary tract infection (Infections and infestations) | 1 | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Splenic injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 1
Adams-Stokes syndrome (Cardiac disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Penile neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 2
Confusional state (Psychiatric disorders) | 0 | 1 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Donepezil + Placebo (N=225) | Donepezil + SB-742457 15 mg (N=221) | Donepezil + SB-742457 35 mg (N=236)
Nasopharyngitis (Infections and infestations) | 17 | 19 | 18
Urinary tract infection (Infections and infestations) | 15 | 10 | 13
Fall (Injury, poisoning and procedural complications) | 12 | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.